CLINICAL TRIAL: NCT06601140
Title: Evaluation of the Concordance Between Measures Obtained by a Medical Device for Emotional Monitoring (EMOCARE) and the Patient Health Questionnaire (PHQ-9) Score in Patients With Mild to Severe Depressive Episode: Prospective, Multicentric, Comparative, Single Blind Clinical Investigation. EMC1 Study
Brief Title: Evaluation of the Concordance Between Measures Obtained by a Medical Device for Emotional Monitoring (EMOCARE) and the Patient Health Questionnaire (PHQ-9) Score in Patients With Mild to Severe Depressive Episode
Acronym: EMC1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emobot (Industry)
Collaborators: Nantes University Hospital (Other); Private psychiatric practice, Saint-Nazaire (Unknown); Groupement Hospitalier Paul Guiraud, Villejuif (Unknown); Centre Hospitalier Guillaume Régnier, RENNES (Unknown); Centre de Psychothérapie Nancéen, Laxou (Unknown); Rumb (Unknown); Private psychiatric pratice, Agen (Unknown); Private psychiatric pratice, Caen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EB-EMC1-2024; 2024-A01487-40 (Other: ANSM)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The participant will continuously use the EMOCARE software during the 6 weeks of follow-up and will answer the questionnaires usually used on a regular basis over the same period.
Masking Description: Patient health questionnaire - 9 (PHQ-9) and (Montgomery Asberg Depression Rating Scale) MADRS assessments will be performed by an investigator who doesn't know the score obtained with EMOCARE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMOCARE (Experimental)
  Interventions: Device: EMOCARE software

INTERVENTIONS:
Device: EMOCARE software — Use of the EMOCARE software on the digital device of participant (smartphone, computer, etc.). The participant can activate and deactivate the software whenever he wishes.

SUMMARY:
The aim of this clinical investigation is to find out whether the EMOCARE emotional monitoring software provides consistent results compared with the tools available for assessing the emotional state of patients suffering from mild to moderately severe depressive episod. It will also provide information on how patients feel about the use of passive monitoring software (without the active involvement of patient). The main questions it aims to answer are as follows:

Does EMOCARE provide consistent results compared with tools already used in current practice? What are the medical problems encountered by participants when using EMOCARE?

The researchers will compare EMCOCARE to various questionnaires usually used in the management of patients suffering from depression (PHQ-9, MADRS, GAD-7, BDI-II, EQ-5D-5L).

Participants who agree to take part in the study, during a selection visit, will be able to:

1. Install the software on a digital interface (smartphone, computer, etc.) and activate or deactivate it whenever they wish during the 6-week follow-up period.
2. Attend 2 scheduled appointments at the centre (a first appointment then a second 6 weeks later) to complete a series of questionnaires, being questioned by the doctor, and fill in other questionnaires on their own.
3. At home, answer questionnaires independently, 2 weeks and 4 weeks after the first appointment.
4. Receive a telephone call from the doctor 3 weeks after the first appointment to find out how the participants are feeling.
5. Keep a diary with the symptoms they have experienced, any medical consultations they have made, or changes in drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes aged 18 or over.
* Outpatient with unipolar depression (regardless of the time of the episode) (major depressive disorder).
* Patient with an episode of major depression supported by PHQ-9 score greater than or equal to 5.
* Patient with an episode of major depression supported by MADRS score greater than or equal to 7.
* Patient accustomed to regular use of a smartphone and/or computer
* Patient who, in the opinion of the investigator, will comply with the requirements of the protocol.
* Patient affiliated to a social security scheme or beneficiary of such a scheme.
* Patient who has received full information about how the clinical investigation shall be conducted and has signed an informed consent form.
* Patient who reads and understands French.
* Patient who has undergone clinical screening adapted to the clinical investigation.

Exclusion Criteria:

* Patient treated with antipsychotic drugs.
* Patient with an unstable pathology that could interfere with the study.
* Patient unable to communicate or cooperate with the investigator due to a low mental level, language difficulties or impaired cerebral function.
* Patient with an active suicidal tendency or patient who has had a suicidal episode in the last 6 months
* Patients with borderline personality disorders.
* Patient with a contra-indication to the product(s) under evaluation.
* Woman of childbearing age without effective contraception.
* Pregnant woman, birthing or breastfeeding mother
* Minor (not emancipated)
* Incapacitated person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-02-04 (Estimated); Study Completion 2027-02-04 (Estimated)

PRIMARY OUTCOMES:
Change of scores EMOCARE | From baseline to 6 weeks
  Absolute difference
Change of scores PHQ-9 self-administrered | From baseline to 6 weeks
  Absolute difference

SECONDARY OUTCOMES:
Score EMOCARE | At baseline, at 2 weeks, at 4 weeks
Change of EMOCARE score | From baseline to 2 weeks, from baseline to 4 weeks
Score PHQ-9 self administered | At baseline, at 2 weeks, at 4 weeks, at 6 weeks
Change of score PHQ-9 self administered | From baseline to 2 weeks, From baseline to 4 weeks
Score PHQ-9 administered by an investigator | At baseline, at 6 weeks
Change of score PHQ-9 administered by an investigator | From baseline to 6 weeks
Score MADRS administered by an investigator | At baseline, at 6 weeks
Change of MADRS administered by an investigator | From baseline to 6 weeks
Score BDI-II | At baseline, at 6 weeks
Change of BDI-II | From baseline to 6 weeks
Score BDI-II | At baseline, at 2 weeks, at 4 weeks, at 6 weeks
Change of BDI-II | From baseline to 2 weeks, from baseline to 4 weeks, from baseline to 6 weeks
EMOCARE operating time | From baseline to 2 weeks, from baseline to 4 weeks, from baseline to 6 weeks
EQ-5D-5L | At baseline, at 6 weeks
Number of patient with adverse event | At baseline, at 2 weeks, at 3 weeks, at 4 weeks, at 6 weeks
Acceptability of medical device questionnaire | At baseline, at 6 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Private psychiatric practice, Agen
  - Private psychiatric pratice, Caen
  - Centre Psychothérapique de Nancy, Laxou
  - Private psychiatric practice, Maxéville
  - Private psychiatric practice, Nantes
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre hospitalier Guillaume Régnier, Rennes
  - Private psychiatric practice, Saint-Grégoire
  - Private psychiatric practice, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No